CLINICAL TRIAL: NCT04906486
Title: Clinical Assessment of Autonomic Functions by SCOPA-Autonomic Questionnaire in Patients With Restless Legs Syndrome: A Prospective Study in a Tertiary Care Hospital
Brief Title: Autonomic Assessment in Patients With Restless Legs Syndrome
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Sehnaz Basaran, Principal Investigator, Department of Neurology, Kocaeli Derince Education and Research Hospital
Other Study IDs: 2011-KAEK-27/2020-E.2000173683
Record Dates: First submitted 2021-05-22; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Restless Legs Syndrome
Keywords: restless legs syndrome; autonomic dysfunction; dysautonomia; SCOPA-AUT questionnaire
MeSH Terms: conditions — Restless Legs Syndrome; Primary Dysautonomias; Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational: Patients with restless legs syndrome: A total of 70 patients who diagnosed with primary restless legs syndrome according to the five essential criteria as established by the International Restless Legs Syndrome Study Group.
- Observational: Healthy controls: The control group consisted of 85 age- and gender-matched healthy volunteers.

SUMMARY:
Restless legs syndrome (RLS) is a sensorimotor, sleep-related disorder characterized by urgency to move the legs during inactivity or resting state. Although the exact mechanism is not clearly understood, sleep disturbances and dopamine deficiency may regarded as a potential contributing factor for autonomic dysfunction. The objective of the study is to evaluate autonomic functions and determine possible associations between autonomic dysfunction with clinical factors in patients with RLS.

DETAILED DESCRIPTION:
Restless legs syndrome (RLS) also known as Willis- Ekbom disease, is a common sensorimotor, sleep-related disorder characterized by an unpleasant feeling with urgency to move the legs (or less commonly the arms) during inactivity or resting state.

Although, the clinical importance of autonomic involvement in patients with restless legs syndrome (RLS) remains incompletely understood, sleep disturbances and dopamine deficiency may regarded as a potential contributing factor for autonomic dysfunction.

Previous reports have described autonomic impairment including changes in nocturnal blood pressure and heart rate variability (HRV), gastrointestinal, urinary and sexual dysfunction in patients with RLS. Despite many studies about electrophysiological autonomic changes in RLS, number of studies exploring autonomic functions by using Scales for Outcomes in Parkinson's disease-Autonomic questionnaire (SCOPA-AUT) are limited.

In this study, the investigators plan to compare the presence of autonomic symptoms by using Scales for Outcomes in Parkinson's disease-Autonomic (SCOPA-AUT) questionnaire in drug- naive RLS patients to healthy controls. In addition, the investigators aim to evaluate possible associations between autonomic dysfunction with clinical factors in patients with RLS.

ELIGIBILITY:
Inclusion Criteria:

For the patient group:

* age >18, <65
* newly diagnosed, drug naive patients with primary restless legs syndrome

For the control group:

* age >18, <65
* participants without chronic systemic disorder

Exclusion Criteria:

* previous diagnosis of primary RLS
* subjects with secondary RLS
* concomitant use of drugs that could interfere with autonomic nervous system
* individuals with a known acute/chronic medical disease
* individuals with a minimental test score < 25/30
* sleep disorders that could affect test performances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were selected from a tertiary care neurology outpatient clinic. Age and gender matched control group obtained from the family members of the tertiary care hospital's staff.
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Scales for Outcomes in Parkinson's disease-Autonomic questionnaire (SCOPA-AUT) (points) | 6 months
  Presence and severity of autonomic dysfunction noted by using Scales for Outcomes in Parkinson's disease-Autonomic questionnaire [SCOPA-AUT, including six domains (gastrointestinal,urinary, cardiovascular, thermoregulatory, pupillomotor, and sexual) with 25-items and a 4 -point Likert-type scale ranging from 0 to 69] in patients with restless legs syndrome vs. healthy controls.
Age (years) | 6 months
  Correlation between autonomic dysfunction and age (years) in patients with restless legs syndrome noted.
Age of disease onset (years) | 6 months
  Correlation between autonomic dysfunction and age of disease onset (years) in patients with restless legs syndrome noted.
Disease duration (years) | 6 months
  Correlation between autonomic dysfunction and disease duration (years) in patients with restless legs syndrome noted.
Disease severity (as measured by International Restless Legs Scale) (points) | 6 months
  Correlation between autonomic dysfunction and disease severity (as measured by International Restless Legs Scale,5-point Likert-type scale ranging from 0 to 40; mild= 0-10; moderate= 11-20; severe= 21-30; very severe= 31-40) in patients with restless legs syndrome noted.
Excessive daytime sleepiness (as measured by Epworth Sleepiness scale) (points) | 6 months
  Correlation between autonomic dysfunction and excessive daytime sleepiness [as measured by Epworth Sleepiness scale ,8-items with a 4-point Likert-type scale ( 0=would never doze,1=slight chance,2=moderate chance, 3= high chance) ranging from 0 to 24 points] in patients with restless legs syndrome noted.
Body mass index (kg/m2) | 6 months
  Correlation between autonomic dysfunction and body mass index (kg/m2, as calculated by dividing weight in kilograms by their height in metres squared) in patients with restless legs syndrome noted.

CONTACTS AND LOCATIONS:
Overall Officials: SEHNAZ BASARAN, MD, Principal Investigator — KOCAELİ DERİNCE EDUCATION AND RESEARCH HOSPİTAL DEPARTMENT OF NEUROLOGY
Locations (1):
- Sehnaz Basaran, İzmit, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet

REFERENCES:
- [Derived] Basaran S, Akinci E. Screening autonomic functions in patients with restless legs syndrome: A case-control study in a tertiary care hospital. Auton Neurosci. 2022 Jan;237:102924. doi: 10.1016/j.autneu.2021.102924. Epub 2021 Nov 29. PMID 34871924